CLINICAL TRIAL: NCT05417815
Title: Interest of Nitazoxanide Treatment of Enterocytozoon Bieneusi Intestinal Microsporidiosis
Acronym: NITAZO-SPORE
Status: Completed | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: 2022 POIRIER NITAZO-SPORE
Record Dates: First submitted 2022-06-02; First posted 2022-06-14 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-05

CONDITIONS: Microsporidiosis Intestinal
Keywords: microsporidia; Enterocytozoon bieneusi; solid organ transplant

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Microsporidia are pathogenic fungi mainly responsible for profuse watery diarrhea, requiring management in immunocompromised patients. The main immunocompromised population affected by these infections consists of solid organ transplant recipients (SOT), mainly kidney (~70% of cases in immunocompromised patients). In this population, the infection is severe, and becomes chronic in the absence of appropriate care, the species Enterocytozoon bieneusi being found in more than 95% of these cases. Reducing immunosuppression (adjustment of immunosuppressive therapy) can sometimes be enough to eliminate the pathogen. However, in some cases, specific treatment is necessary. The only molecule whose efficacy has been proven to date to treat infections caused by E. bieneusi is fumagillin (FLISINT®), however its production has been stopped for almost 2 years. Due to the therapeutic impasse, the use of nitazoxanide (ALINIA®) to treat E. bieneusi microsporidiosis is becoming common, despite the lack of proof of its efficacy. It seems important and urgent to evaluate the relevance of the use of nitazoxanide, particularly in SOT, for the treatment of intestinal microsporidiosis due to E. bieneusi.

ELIGIBILITY:
Inclusion Criteria:

* With a diagnosis of intestinal infection caused by E. bieneusi between 01/01/2018 and 03/31/2022
* having received treatment with nitazoxanide ("NITAZO" group), or fumagillin ("FUMA" group), or albendazole ("ABZ") or having received no specific treatment but having benefited from an adjustment of the doses of immunosuppressants ("IS" group)

Exclusion Criteria:

* With a diagnosis of extraintestinal infection
* With a diagnosis of infection by a species other than E. bieneusi

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: SOT with microsporidiosis
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
efficiency by symptoms | 1 year
  time to resolution of symptoms
efficiency by parasitology | 1 year
  parasitological negativation
efficiency by relapses | 1 year
  number of relapses
tolerance of treatment | 1 year
  duration of treatment
tolerance with side effects | 1 year
  side effects during treatment: value of platelets, liver enzymes, occurrence of drug interactions

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Poirier, Study Director — University Hospital, Clermont-Ferrand
Locations (24):
- France (23):
  - CHU Amiens, Amiens
  - CHU Besançon, Besançon
  - CHU Bordeaux, Bordeaux
  - CHU Brest, Brest
  - CHU Caen, Caen
  - CHU clermont-ferrand, Clermont-Ferrand
  - CHU Dijon, Dijon
  - CHU Grenoble, Grenoble
  - CHU Lille, Lille
  - CHU Limoges, Limoges
  - Hospices Civils de Lyon, Lyon
  - AP-HM, Marseille
  - CHU Nancy, Nancy
  - AP-HP Hopital Bichat Claude-Bernard, Paris
  - AP-HP Hopital Necker-Enfants Malades, Paris
  - AP-HP Hopital Saint-Antoine, Paris
  - AP-HP Hopitaux Universitaires Henri-Mondor, Paris
  - CHU Poitiers, Poitiers
  - CHU Rouen, Rouen
  - CHU Saint-Etienne, Saint-Etienne
  - CHU Strasbourg, Strasbourg
  - CHU Toulouse, Toulouse
  - CHU Tours, Tours
- CHU Pointe-à-Pitre, Pointe-à-Pitre, Guadeloupe

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Garrouste C, Poirier P, Uro-Coste C, Iriart X, Kamar N, Bonhomme J, Calvar E, Le Gal S, Lanfranco L, Autier B, Rakoff L, Durieux MF, Danthu C, Morio F, Deltombe C, Moreno-Sabater A, Ouali N, Costa D, Bertrand D, Chesnay A, Gatault P, Rabodonirina M, Morelon E, Dumortier J, Sitterle E, Scemla A, Hamane S, Cachera L, Damiani C, Poulain C, L'Ollivier C, Moal V, Delhaes L, Kaminski H, Cateau E, Ecotiere L, Brunet J, Caillard S, Valot S, Tinel C, Argy N, Raimbourg Q, Robert MG, Noble J, Boignard A, Botterel F, Matignon M, Bellanger AP, Crepin T, Leroy J, Lionet A, Debourgogne A, Nicolas M, Claudeon J, Moniot M, Lambert C, Nourrisson C. Fumagillin Shortage: How to Treat Enterocytozoon bieneusi Microsporidiosis in Solid Organ Transplant Recipients in 2024? Transpl Int. 2024 Dec 12;37:13518. doi: 10.3389/ti.2024.13518. eCollection 2024. PMID 39726674